CLINICAL TRIAL: NCT04175652
Title: Effects of Laughter Yoga on Hemodialysis Patients' Plasma-Beta Endorphin Levels, Pain Levels and Sleep Quality: A Randomized Controlled Trial
Brief Title: Effects of Laughter Yoga on Hemodialysis Patients' Plasma-Beta Endorphin Levels, Pain Levels and Sleep Quality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Sabahattin Zaim University (Other)
Responsible Party: Principal Investigator, Zülfünaz ÖZER, PhD., Assistant Prof., Istanbul Sabahattin Zaim University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2017-314
Record Dates: First submitted 2019-11-21; First posted 2019-11-25 (Actual); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Laughter Yoga; Hemodialysis Patients
Keywords: Laughter Yoga; Hemodialysis; Pain; Sleep; Beta Endorphin
MeSH Terms: conditions — Pain | interventions — Laughter Therapy

STUDY DESIGN:
Intervention Model Description: Parallel Assignment Randomization; participants were divided into two groups by using simple random numbers table, and then the first group which was drawn by lot method was named as the experimental group.
Who Masked: Investigator
Masking Description: Single
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laughter yoga group, group doing laughter yoga (Experimental): The duration of the laughter yoga was 30 minutes and a total of 16 sessions were performed on a twice-weekly basis.
  Interventions: Behavioral: Laughter yoga
- No laughter yoga group, group not doing laughter yoga (No Intervention)

INTERVENTIONS:
Behavioral: Laughter yoga — The laughter yoga practice was initiated through clapping and warm-up exercises: hands were clapped keeping hands in parallel with each other and ensuring that the fingertips touched each other. To increase the energy level of the group, a rhythmic beat was added to the clapping in the form of 1-2, 1-2-3. While this was being sung a rhythm was tapped out on the floor by moving the feet up and down. Eye contact was constantly maintained with the participants. In the second phase, deep breathing exercises were performed. Participants were encouraged to inhale from the diaphragm. Individuals were asked to put their hands on their belly and inhale through the nose and then slowly exhale through the mouth. After the deep breathing exercise, the participants were encouraged to laugh through playing children's games in the third phase.
  Arms: Laughter yoga group, group doing laughter yoga

SUMMARY:
This study aimed to assess the effectiveness of laughter yoga on HD patients' plasma beta endorphin levels, pain levels and sleep quality.

DETAILED DESCRIPTION:
While there are studies conducted with laughter yoga on different patient groups in Turkey, no studies have been found on hemodialysis patients specifically. For this reason, it was thought that studies are needed which will prove the effect of laughter yoga practices on the plasma beta-endorphin levels, pain levels and sleep quality of hemodialysis patients.

ELIGIBILITY:
Inclusion Criteria:

* receiving treatment in a dialysis center
* must be between 18 and 80 years old and willing to participate in the study
* receiving HD treatment at least twice a week for a month or longer
* having a pain level and above
* level of 5 above according to the Pittsburgh Sleep Quality Index.

Exclusion Criteria:

* not taking any medicine for sleeping disorder
* not having any visual, hearing or communication impairments
* not having any mental disorders

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2017-11-15 (Actual); Primary Completion 2018-06-15 (Actual); Study Completion 2018-10-31 (Actual)

PRIMARY OUTCOMES:
Beta-endorphin Level | 8 week
  Blood samples were taken from all individuals who participated in the study, through their AVF fistulas by using 3.5 mL gel-based tubes and following antiseptic rules. Blood samples which were fully coagulated were centrifuged at 1500xg for 10 minutes and serums were obtained. The serum samples were separated into portions and kept at -80 °C until the analysis.
Visual Analog Scale | 8 week
  The patients were asked to mark their level of pain during relaxation or activities on a 10 cm vertical or horizontal line. In addition, there were forms which were numbered from 1-10 or from 1-100. The number 0 is found at the beginning of the line, and the number 10 is located at the end of the line. A value of 0 shows that there is no pain, and the value 10 expresses unendurable pain. GAS is a common scale in the assessment of pain level. A patient is asked to mark the perceived pain on this line, and the marked point is measured in cm
Pittsburgh Sleep Quality Index | 8 week
  The PSQI is a valid and consistent survey comprising of 19 questions to assess quality and amount of sleep and the existence of a sleep disorder and its level in the previous month. The scale was adapted into the Turkish language by Agargün et al. (1996). The scale consists of seven components that assess patients subjective sleep quality, sleep delay, use of sleeping medication and disfunction in daily activities. Each item scores in the range 0-3 points and the total score of the seven components gives the total PSQI score. The total score has a value between 0-21 and a high total score demonstrates a poor quality of sleep. A total PSQI score which is ≤5 indicates "good sleep", and a score which is >5 indicates "poor sleep"

CONTACTS AND LOCATIONS:
Overall Officials: Zülfünaz Ozer, Dr, Principal Investigator — Istanbul Sabahattin Zaim University
Locations (1):
- Istanbul Sabahattin Zaim University, Faculty of Health Sciences, Istanbul, Küçükçekmece, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
after the article is published

REFERENCES:
- [Background] Heo EH, Kim S, Park HJ, Kil SY. The effects of a simulated laughter programme on mood, cortisol levels, and health-related quality of life among haemodialysis patients. Complement Ther Clin Pract. 2016 Nov;25:1-7. doi: 10.1016/j.ctcp.2016.07.001. Epub 2016 Jul 27. PMID 27863598
- [Background] Yim J. Therapeutic Benefits of Laughter in Mental Health: A Theoretical Review. Tohoku J Exp Med. 2016 Jul;239(3):243-9. doi: 10.1620/tjem.239.243. PMID 27439375